CLINICAL TRIAL: NCT01138943
Title: Chlorhexidine Alcohol Base Mouthrinse Versus Chlorhexidine Formaldehyde Base Mouthrinse Efficacy on Plaque Control: Double Blind, Randomized Clinical Trials
Brief Title: Chlorhexidine Mouthrinses and Plaque Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Militaire De Rabat (Other)
Collaborators: CCTD, Centre Hospitalier Ibn Sina,Morocco (Unknown); Faculté de Médecine Dentaire de Rabat (Unknown); Faculté de Médecine de Rabat (Unknown); Mohammed V Souissi University (Other)
Responsible Party: Ennibi Oumkeltoum , Head of clinical Department of Periodontology, Faculté de Médecine Dentaire de Rabat
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1251/10; 1171 (Other: Comité d'Ethique de la Recherche Biomédicale (CERB))
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2007-02

CONDITIONS: Dental Plaque
Keywords: Chlorhexidine mouthrinse; Plaque control
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine alcohol-base mouthrinse (Active Comparator)
  Interventions: Drug: Synthodont
- non alcohol chlorhexidine mouthrinse (Experimental)
  Interventions: Drug: Soludent

INTERVENTIONS:
Drug: Synthodont — 15 ml, tree times/day for 07 days
  Arm: Chlorhexidine alcohol-base mouthrinse
  Arms: Chlorhexidine alcohol-base mouthrinse
Drug: Soludent — 15ml of 01% Chlorhexidine non alcohol-based, 3 times a day for 7 days
  Arm: Experimental: non alcohol chlorhexidine mouthrinse
  Arms: non alcohol chlorhexidine mouthrinse

SUMMARY:
The aim of the present study was to compare antiplaque effectiveness of two commercial mouthrinses: 0.12 % Chlorhexidine alcohol base (CLX-A) versus a diluted 0.1% Chlorhexidine non-alcohol base with 0.1% of Formaldehyde (CLX-F).

DETAILED DESCRIPTION:
Chlorhexidine (CLX) mouthrinse has been the gold standard as antiplaque solution.However, if its efficiency seems to be preserved even if the chlorhexidine concentration is bellow 0.10%, the formulation of the final product may affect the effectiveness. Thus, it can be concluded from this study that 0.12% CLX alcohol base mouthrinse is significantly more effective in inhibiting plaque than the diluted 0.1% CLX non-alcohol base containing formaldehyde mouthrinse.

ELIGIBILITY:
Inclusion Criteria:

* give written informed consent before entering the study
* accept to stop tooth cleaning for a week

Exclusion Criteria:

* less than 20 teeth;
* presence of periodontal disease
* presence of factors of plaque retention (clinically unacceptable restorations, important carious, dental overlapping, removable prosthesis, faulty fixed prosthesis, orthodontic appliances),
* associated systemic diseases (diabetes, heart disorders, blood diseases, HIV infection),
* use of antibiotics or other anti-inflammatory drugs during the latest months,
* known allergy against components of mouth rinses,
* pregnancy,
* smoking

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Plaque Index (PI)at Day 1 and Day 7. | one week
  The clinical trial lasted 7 days (from Day 0 to Day 7). During this period all participants abstained from all mechanical oral hygiene procedures.
  On Day 0, subjects were randomly distributed in three groups: two test groups and one negative control group, and were instructed to rinse twice daily with the allocated mouthrinse during the experimental period.
  The clinical measurement: Plaque Index (PI) was recorded on Day 1 and Day 7.

SECONDARY OUTCOMES:
Side effects | at day 7
  On Day 7, all subjects were examined for the presence or absence of tooth staining, and were questioned about taste disturbances and mucosal sensitivities.

CONTACTS AND LOCATIONS:
Overall Officials: Oumkeltoum Ennibi, Professor, Study Chair — Faculté de Médecine Dentaire
Locations (1):
- Faculté de Médecine Dentaire, Rabat, Morocco